CLINICAL TRIAL: NCT00541840
Title: Phase I-II, Not-Randomized, Multicenter Clinical Trial to Evaluate Safety and Efficacy of Sorafenib (BAY-43-9006) in Combination With Ifosfamide in Soft Tissue Sarcoma.
Brief Title: Phase I-II Trial of Sorafenib in Combination With Ifosfamide in Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Grupo Espanol de Investigacion en Sarcoma, Grupo GEIS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS01-07
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Soft Tissue Sarcoma
Keywords: Sarcoma; Sorafenib; GEIS
MeSH Terms: conditions — Sarcoma | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sorafenib — Phase I:
  Level 1: Sorafenib 200 mg bid, orally Ifosfamide 2,0 g/m2, intravenously, over 4 hours, on 3 consecutive days Mesna 400 mg/m2 iv, at 0, 4 and 8 hours after the Ifosfamide administration
  Level 2: Sorafenib 400 mg bid, orally Ifosfamide 2.00 g/m2, intravenously, over 4 hours, on 3 consecutive days Mesna 400 mg/m2 iv, at 0, 4 and 8 hours after the Ifosfamide administration
  Level 3 : Sorafenib 400mg bid, orally Ifosfamide 2.5 g/m2 , intravenously , over 4 hours , on 3 consecutive days . Mesna 500mg/m2,iv,at 0,4 and 8 hours after ifosfamide administration .
  Level 4 : Sorafenib 400 mg bid, orally Ifosfamide 3.0 g/m2, intravenously, over 4 hours, on 3 consecutive days Mesna 600 mg/m2 iv, at 0, 4 and 8 hours after the Ifosfamide administration
  Phase II:
  Sorafenib and Ifosfamide administered at the doses recommended in phase I until progression or unacceptable toxicity.
  Other Names: BAY 43-9006

SUMMARY:
Soft tissue sarcomas (STS) are an uncommon group of malignant tumors of mesenchymal origin. For most advanced STS types, chemotherapy is currently the only available treatment. Unfortunately, a very limited number of useful drugs are active against this disease. Doxorubicin is widely considered the standard first-line treatment. Ifosfamide has also a well-established activity (1,2) and is often administered either associated with Doxorubicin or alone as a second-line chemotherapy treatment. Other drugs such as DTIC, Gemcitabine and Temozolomide showed modest activity as a second-line agents (3,4). Thus, there is a necessity to identify new agents with activity to improve therapy for patients with advanced STS. In some studies, most STS showed VEGF expression, and elevated serum VEGF levels were found to correlate with higher histologic tumor grade (5,6). Additionally, inhibition of VEGFR was associated with tumor activity in preclinical models of sarcoma (7,8). For these reasons, inhibition of VEGFR seems to be a reasonable approach to explore in the treatment of STS. Sorafenib (BAY 43-9006) is an orally available, small molecule multi-kinase inhibitor of VEGFR, PDGFR and RAF with demonstrated activity in the treatment of renal cell cancer (9). Preclinical studies suggest that the combination of Sorafenib with cytotoxic agents results in additive anti-tumor activity (10), initiating justification for combination studies. A recent trial, however, reported an unexpected incidence of cardiac toxicity in patients with STS treated with Bevacizumab, a monoclonal antibody that binds VEGF, in combination with Doxorubicin (11). This finding suggest that the possibility of potentiation of the cardiotoxicity of Doxorubicin when inhibiting the VEGF pathway cannot be ruled out. The association of Sorafenib with Ifosfamide, the other established active agent against STS, could improve the efficacy of single-agent Ifosfamide minimizing the risk of cardiac toxicity .

ELIGIBILITY:
Inclusion Criteria:

1. Advanced Soft Tissue Sarcoma histologically proven, excluding the following subtypes: chondrosarcoma, osteosarcoma, Ewing's sarcoma, and embryonal rhabdomyosarcoma.
2. Patients must have been previously treated with Anthracycline. However, patients not eligible for Anthracycline treatment can be included.Prior treatment with Ifosfamide is not allowed, except if it was administered as adjuvant therapy.
3. Patients must be > 18 and < 72 years old.
4. Patients must have ECOG performance status 0 to 1 on fase I.
5. Patients must have ECOG performance status 0 to 2 on fase II.
6. Patients must have measurable disease. Progression must be documented during the last month pre-study entry. No prior radiotherapy in the indicator lesion is allowed.
7. Adequate bone marrow, renal and hepatic function

   * hemoglobin ³ 9.0 g/dl
   * absolute neutrophil count ³ 1,500/mm3
   * platelet count ³ 100,000/mm3
   * total bilirubin £ 1.5 times the upper limit of normal
   * ALT and AST £ 2.5 times the upper limit of normal (£ 5 x upper limit of normal for patients with liver involvement)
   * INR £ 1.5 and aPTT within normal limits
   * serum creatinine £ 1.5 the upper limit of normal
8. Signed informed consent prior to any study specific procedures

Exclusion Criteria:

1. Patients with previous chemotherapy or radiotherapy, within 3 weeks prior to study entry.
2. Pregnant or breast feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days prior to the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
3. Life expectancy of less than 12 weeks.
4. General medical or psychological conditions that would preclude appropriate informed consent or compliance with the protocol.
5. Substance abuse, medical, psychological or social conditions that may interfere with the patients participation in the study.
6. Previous cancer that is distinct in primary site or histology from NSCLC except cervical cancer in-situ, treated basal cell carcinoma, superficial bladder tumors (Ta and Tis) or any cancer curatively treated > 3 years prior to study entry.
7. Concurrent treatment with other anti-cancer therapy.
8. Concurrent treatment with other experimental drugs (within 30 days prior to study entry).
9. Significant weight loss (> or equal 10% body weight during preceding 6 weeks).
10. Major surgery, open biopsy or significant traumatic injury within 4 weeks of first dose of study drug.
11. Biological modifying agents such as G-CSF administered within 3 weeks prior to study entry.
12. Known or suspected allergy to sorafenib or ifosfamide.
13. Evidence or history of bleeding diathesis or coagulopathy.
14. Therapeutic anticoagulation with Vitamin K antagonists such as warfarin or with heparins or heparinoids. Low dose warfarin is permitted if INR is <1.5. Low dose aspirin is permitted.
15. Thrombotic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months.
16. Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal medical management.
17. Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina or new-onset angina (began within the last 3 months) or myocardial infarction within the last 6 months.
18. Active clinically serious infections > CTCAE Grade 2.
19. Serious, non-healing wound, ulcer, or bone fracture.
20. Concomitant treatment with ketoconazole, itraconazole, ritonavir, rifampicin and St. John´s Wort.
21. Known HIV infection or chronic hepatitis B or C.
22. Known brain metastasis. Patients with neurological symptoms should undergo a CT scan/MRI of the brain to exclude brain metastasis.
23. Any other condition that could compromise patient's security and/or study's fulfilment.
24. Known or suspected allergy to mesna or tiolic agents.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Phase I: Safety profile and to determine maximum tolerated dose (MTD) / Recommended Dose (DR) of Sorafenib in combination with Ifosfamide. Phase II: Activity profile evaluating of the combination in patients with advanced soft tissue sarcoma. | Phase II: Progression free rate: at 3 and 6 months

SECONDARY OUTCOMES:
Phase II: Efficacy evaluation | Phase II: Progression free rate at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Garcia del Muro, MD, Study Director — Grupo Español de Investigacion en Sarcomas (GEIS)
Locations (1):
- Grupo Geis, Madrid, Madrid, Spain

REFERENCES:
- See also: Grupo Español de Investigacion en Sarcomas Website — http://www.grupogeis.org/